CLINICAL TRIAL: NCT06565286
Title: Inlay Inner Preputial Graft Versus Transverse Preputial Island Flap in Management of Proximal Penile Hypospadias
Brief Title: Graft Versus Flap in Management of Proximal Penile Hypospadias
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Shabaan Abohamady, assistant lecturer- urology departement - faculty of medicine -sohag university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-24-06-02MD
Record Dates: First submitted 2024-08-11; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Proximal Penile Hypospadias

STUDY DESIGN:
Intervention Model Description: Inlay inner preputial graft versus Transverse preputial island flap in management of proximal penile hypospadias
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inner preputial graft (Active Comparator): managemet of proximal penile hypospadias in 2stage using inner preputial graft in the first stage
  Interventions: Procedure: inner preputial graft versus transverse preputial island flap in two-stage repair of proximal penile hypospadias
- transverse preputial island flap (Active Comparator): managemet of proximal penile hypospadias in 2stage using transverse preputial island flap in the first stage
  Interventions: Procedure: inner preputial graft versus transverse preputial island flap in two-stage repair of proximal penile hypospadias

INTERVENTIONS:
Procedure: inner preputial graft versus transverse preputial island flap in two-stage repair of proximal penile hypospadias — compare outcomes of inner preputial graft versus transverse preputial island flap when used to substitute the urethral plate in two-stage repair of primary proximal penile hypospadias .
  Other Names: graft versus flap in two-stage repair of proximal penile hypospadias

SUMMARY:
Proximal hypospadias (penoscrotal, scrotal, and perineal types) account for approximately 20% of all cases . The management of hypospadias has greatly improved over the past two decades since the introduction of tubularized incisized plate urethroplasty. However, obtaining a favorable cosmetic outcome and functional straight penis is a major surgical challenge for such patients, and the ideal repair of proximal hypospadias remains the Holy Grail for hypospadias specialists.

DETAILED DESCRIPTION:
The surgical plan for proximal hypospadias can be divided into single and staged operations. Single stage operations are often associated with high rates of complications and reoperations. Reportedly, complications occur in 20-50% of patients. Therefore, many pediatric surgeons are selecting staged procedures. Staged surgical repair of proximal forms of hypospadias has been proven to achieve successful both functional and cosmetic results. Although staged repair with inner preputial layer graft has regained popularity in the repair of proximal hypospadias; but Choosing between flaps or grafts to substitute the urethral plate in 2-stage hypospadias repair has been a matter of debate with no consensus in the literature.

Flaps have reliable blood supply that may be theoretically less liable for strictures or contractures. Grafts are more versatile, which can be used in primary and recurrent cases when healthy local skin is deficient.

In this study, our aim is to compare outcomes of grafts and flaps when used to substitute the urethral plate in two-stage repair of primary proximal penile hypospadias (penoscrotal and scrotal types).

ELIGIBILITY:
Inclusion Criteria:

* Age: more than 6 months.
* Type of hypospadias: proximal penile hypospadias (scrotal and penoscrotal variants)

Exclusion Criteria:

* Age: less than 6 months.
* Perineal hypospadias.
* circumcised patients.
* Previous hypospadias repair
* Raised serum creatinine, coagulopathy.

Min Age: 6 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — outcomes of graft versus flap in management of proximal penile hypospadius
Enrollment: 50 (Estimated)
Dates: Start 2024-08-18 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
measure complications after staged repair of proximal penile hypospadias using different techniques. | 6 month after end of treatment
  urinary fistulas, urethral strictures, diverticula and failed repair.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed diaa, professor, Study Director — Sohag University
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
Report the cosmotic and functional outcomes after staged repair of proximal penile hypospadias using different techniques.

REFERENCES:
- [Result] Kojima Y, Kohri K, Hayashi Y. Genetic pathway of external genitalia formation and molecular etiology of hypospadias. J Pediatr Urol. 2010 Aug;6(4):346-54. doi: 10.1016/j.jpurol.2009.11.007. Epub 2009 Dec 7. PMID 19995686
- [Result] Bouty A, Ayers KL, Pask A, Heloury Y, Sinclair AH. The Genetic and Environmental Factors Underlying Hypospadias. Sex Dev. 2015;9(5):239-259. doi: 10.1159/000441988. Epub 2015 Nov 28. PMID 26613581
- [Result] Hsieh MH, Breyer BN, Eisenberg ML, Baskin LS. Associations among hypospadias, cryptorchidism, anogenital distance, and endocrine disruption. Curr Urol Rep. 2008 Mar;9(2):137-42. doi: 10.1007/s11934-008-0025-0. PMID 18419998
- See also: Genetic pathway of external genitalia formation and molecular etiology of hypospadias — http://pubmed.ncbi.nlm.nih.gov/19995686/
- See also: The Genetic and Environmental Factors Underlying Hypospadias — http://pubmed.ncbi.nlm.nih.gov/26613581/
- See also: Associations among hypospadias, cryptorchidism, anogenital distance, and endocrine disruption — http://pubmed.ncbi.nlm.nih.gov/18419998/